Protocol Number:

Version and Date Received:

# **Cover Page for Informed Consent Form**

Official Study Title: What makes people better at describing photographs?

NCT05444114

Document Date 5/30/24

 Version Date: 3.15.2022

# University of Colorado Colorado Springs (UCCS) Consent to be a Research Subject

<u>Title</u>: What makes people better at describing photographs?

**Principal Investigator**: Lori James, PhD

Funding Source: National Institutes of Health

Key Information You are being asked to choose whether or not you would like to participate in a research study. This study is being conducted to learn more about how various personal and situational characteristics are related to the ability to verbally describe the contents of photographs. Over a videoconference call, you will do an exercise involving a 10-minute audio clip, and then be shown photos and asked to provide detailed descriptions of their content. You will also complete some other surveys and measures via Qualtrics. Participation will take approximately 40-60 minutes. There are minimal risks involved in this study, but you may feel frustrated by the description task or you might become bored with audio clip exercise or the surveys. Collected data will be stored by an identification code, not your name. You will not directly benefit from this study, but it will give researchers a better understanding of how individuals' personality and cognitive traits and setting in which the description task occurs correspond with their ability to produce detailed descriptions.

#### Introduction

You are being asked to be in a research study. This form is designed to tell you everything you need to think about before you decide to consent (agree) to be in the study or not to be in the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study.

Before making your decision:

- Please carefully read this form or have it read to you.
- Please ask questions about anything that is not clear.

Feel free to take your time thinking about whether you would like to participate. By agreeing to be in the study you will not give up any legal rights. You may want to print a copy of the consent form for your records.

<u>Study Overview</u> This study is being conducted to learn more about how various personal and situational factors relate to the ability to describe the content of photographs. Results will be presented as group averages, not as individual responses. Findings may be published in journal articles and presented at conferences.

<u>Procedures</u> You are being asked to be in this research study because you are 18-35 or 60-80 years of age and a native, fluent speaker of American English. First, you will do an exercise involving a 10 minute audio clip, following which you will be asked to describe in detail the contents of 3 photographs for 30-60 seconds each. We will audio record the description task for later transcription and scoring, but your name will not be on the recording. People over age 60 will complete one additional cognitive measure. Everyone will also complete several measures about your cognitive and personality factors on Qualtrics. The entire procedure will take approximately 40-60 minutes to complete.

Other people in this study: Approximately 200 people will participate in this study.

<u>Risks and Discomforts</u> There is minimal risk involved in this study. You might feel frustrated by the description task, or you might become bored while doing the exercise with the audio clip or while completing the surveys. This discomfort is

 Version Date: 3.15.2022

Protocol Number:

Version and Date Received:

not expected to be greater than that experienced during everyday life. You may stop participating in the study at any time without any negative consequences.

<u>Benefits</u> You will not directly benefit from this study, but it will give researchers a better understanding of how individuals' personal traits and situational factors relate to the ability to produce descriptions of photographs.

<u>Compensation</u> UCCS student participants are compensated with 2 SONA system credits. Non-student participants are compensated with a \$15 electronic gift certificate.

### Confidentiality

None of your data will have your name attached to it, nor will the audio recording. Participant information will be kept separately from data, in a secure location. Participant information and data will be stored only by a meaningless participant identification code. Only Dr. James and her research assistants will have access to raw or coded data. All electronic data files will be kept on password-protected computers.

Your confidentiality will be maintained to the degree permitted by the technology used. Specifically, no guarantees can be made regarding the interception of data sent via the Internet by any third parties.

Certain offices and people other than the researchers may have access to study records. Government agencies and UCCS employees overseeing proper study conduct may look at your study records. These offices include the UCCS Institutional Review Board, and the UCCS Office of Sponsored Programs and Research Integrity. UCCS will keep any research records confidential to the extent allowed by law. A participant identification code rather than your name will be used on study records wherever possible. Study records may be subject to disclosure pursuant to a court order, subpoena, law or regulation.

Additionally, there may be instances where the researcher(s) cannot keep information you provide them confidential, including reports of abuse or neglect of a child, at-risk adult, dependent adult, or elder. If such information is reported to the researcher(s), they may have to report it to the appropriate authorities.

If you would like to report an incident, please contact the Office of Institutional Equity at 719-255-4324 or via email equity@uccs.edu or for additional resources visit their website https://equity.uccs.edu/

Your de-identified data collected during this study could be used for future research studies without additional consent. Also, your de-identified data may be made available to the scientific community in an online format as required by sponsors or publishers.

#### **Voluntary Participation and Withdrawal from the Study**

Taking part in this study is voluntary. You have the right to leave the study at any time without penalty. You may refuse to answer any questions that you do not wish to answer. If you withdraw from the study, you may request that your data not be used by contacting the Principal Investigator listed above and below. If you are a UCCS student, there are alternative options to earn credit other than participating in this study. Contact your course instructor if you would like to learn about alternatives for receiving extra credit.

## **Contact Information**

Contact (PI's info): Contact (PI's info): Lori James at ljames@uccs.edu

- if you have any questions about this study or your part in it,
- if you have guestions, concerns or complaints about the research, or
- if you would like information about the survey results when they are prepared.

 Version Date: 3.15.2022

Protocol Number:

Version and Date Received:

Contact the Research Integrity Compliance Program Director at 719-255-3903 or via email at <a href="mailto:irb@uccs.edu">irb@uccs.edu</a>:

- if you have questions about your rights as a research participant, or
- if you have questions, concerns or complaints about the research.

### **Electronic Consent**

Please print a copy of this consent form for your records, if you so desire.

I have read and understand the above consent form, I certify that I am 18 years old or older and, by clicking the submit button to enter the survey, I indicate my willingness to voluntarily take part in the study.

 Version Date: 3.15.2022